CLINICAL TRIAL: NCT01720368
Title: IBD-OPERA Database IBD OPERA Database: Inflammatory Bowel Disease - Outcomes, Preferences, Education, Resource Utilization, Assessment Database - Crohn's Protocol
Brief Title: OPERA Database - Crohn's Protocol
Acronym: OPERA
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: IMM 10-0162
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Inflammatory Bowel Disease; Crohn's Disease
Keywords: IBD; Crohn's
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1st Group of 50 patients
- 2nd Group of 50 patients

SUMMARY:
The investigators believe that patients with Crohn's disease are able to report details of their own medical history accurately and record changes in clinical status effectively over time. Using an internet-based database the investigators will ask patients to report their own disease history, and the investigators will compare their reports to the medical record.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years of age) with physician diagnosed Crohn's disease
* A current or past prescription of anti-TNF
* Access to medical record for validation of clinical information

Exclusion Criteria:

* Unwilling or unable to provide informed consent for study participation
* Unable to access or use the internet
* Ulcerative colitis or IBD-U
* Illiterate or does not possess minimum level of literacy required to complete questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women over 18 years of age with Crohn's disease
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Validity of patient self reporting | 12 months
  The validity of patient self report on details of their Crohn's disease compared to chart review. Validity is defined as a match between patient self report and medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States